# **Statistical Analysis Plan Amendment 1**

Study ID: 209012 Substudy 2

**Sub-study Official Title:** Assessment of Safety and Recommended Phase 2 Dose of Autologous T cells Engineered with an Affinity-enhanced TCR Targeting NY-ESO-1 and LAGE-1a, and co-expressing the dnTGF-βRII (GSK3845097) in Participants with NY-ESO-1 and/or LAGE-1a Positive Previously Treated Advanced (Metastatic or Unresectable) Synovial Sarcoma and Myxoid/Round Cell Liposarcoma

NCT ID for sub-study: NCT05943990

**Date of Document:** 03-APR-2023

**Information Type:** Statistical Analysis Plan (SAP)



### TITLE PAGE

**Protocol Title:** Master Protocol to Assess the Safety and Recommended Phase

2 Dose of Next Generations of Autologous Enhanced NY-ESO-1/ LAGE-1a TCR Engineered T cells, alone or in

combination with other agents, in Participants with Advanced

**Tumors** 

**Substudy Title:** Assessment of Safety and Recommended Phase 2 Dose of

Autologous T cells Engineered with an Affinity-enhanced TCR Targeting NY-ESO-1 and LAGE-1a, and co-expressing the dnTGF-βRII (GSK3845097) in Participants with NY-ESO-1 and/or LAGE-1a Positive Previously Treated Advanced (Metastatic or Unresectable) Synovial Sarcoma and

Myxoid/Round Cell Liposarcoma

Study Number: 209012

Compound Number: GSK3845097

**Abbreviated Title:** Substudy 2: GSK3845097 in previously treated advanced

synovial sarcoma and myxoid/round cell liposarcoma

Sponsor Name: GlaxoSmithKline Research & Development Limited

**Regulatory Agency Identifier Number(s)** 

**Registry** ID

IND Number 19751

EudraCT Number 2019-004446-14

Clinicaltrials.gov NCT04526509

Copyright 2023 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | PAGE |
|----|------|-------------------------------------------------|------|
| 1. | INTR | ODUCTION | 5 |
| | 1.1. | Objectives, Estimands, and Endpoints | 5 |
| | | 1.1.1. Objectives and Endpoints | |
| | 1.2. | Study Design | |
| 2. | STAT | FISTICAL HYPOTHESES | 12 |
| | 2.1. | Multiplicity Adjustment | 12 |
| 3. | ANAL | LYSIS SETS | 13 |
| 4. | STAT | ΓISTICAL ANALYSES | 14 |
| | 4.1. | General Considerations | 14 |
| | | 4.1.1. General Methodology | 14 |
| | | 4.1.2. Baseline Definition | |
| | 4.2. | Primary Endpoint(s) Analyses | 14 |
| | 4.3. | Secondary Endpoint(s) Analyses | |
| | 4.4. | Exploratory Endpoint(s) Analyses | |
| | 4.5. | Safety Analyses | |
| | 4.6. | Other Analyses | 15 |
| | | 4.6.1. Subgroup analyses | |
| | 4.7. | 4.7. Interim Analyses | |
| | | 4.7.1. Dose Confirmation Phase | 15 |
| | | 4.7.2. Dose Expansion Phase | 17 |
| | | 4.7.3. Primary Analysis | 17 |
| | | 4.7.4. Final Analysis | |
| | 4.8. | Changes to Protocol Defined Analyses | 18 |
| 5. | SAMI | PLE SIZE DETERMINATION | 19 |
| 6. | SUPF | PORTING DOCUMENTATION | 20 |
| | 6.1. | Appendix 1 Study Population Analyses | |
| | | 6.1.1. Demographic and Baseline Characteristics | 20 |
| 7 | RFFF | FRENCES | 21 |

# **Version history**

| SAP<br>Version | Approval Date Approval Date On which SAP is Based Change | | Rationale | |
|---|---|---|---|---|
| SAP v1 | 17 May 2022 | 209012/Amend<br>ment 3 (20-Dec-<br>2021) | Not Applicable | Original version |
| SAP<br>Amendment<br>1 | 03 Apr 2023 | 209012/Amend<br>ment 4 (27-<br>May-2022) | In addition to minor typographical and formatting changes, the following updates have been made in relation to the reduction in scope of original planned analyses as a result of substudy termination: • Removal of references to summaries based on RP2D or the Evaluable Analysis Set (througho ut document) • Clarificati on on the presentati on of the safety and efficacy analyses | |

| SAP<br>Version | Approval Date | Protocol Version (Date) on which SAP is Based | Change | Rationale |
|---|---|---|---|---|
| | | | (Section 4.1.1) Removal of subgroup analyses (Section 4.6.1) Clarificati on that the protocolplanned Interim and Primary analyses will not be conducted (Section 4.7). Removal of Explorator y colplanted in the core SAP (Section 4.4) | |

# 1. INTRODUCTION

The purpose of this Statistical Analysis Plan (SAP) is to describe the planned analyses to be included in the CSR for Sub-study 2 (GSK3845097) 209012. The core SAP covers the majority of the analyses for this substudy. However, additional details that are specific to this substudy are provided below.

As described in Core SAP Amendment 2, due to early termination of all substudies only a subset of the previously planned analyses are now required. The following key changes to previously planned analyses are relevant to this document: 1) since the substudy was terminated prior to the establishment of the recommended phase 2 dose (RP2D), no related analyses will be provided (e.g., analyses based on the Evaluable analysis set). 2) The Interim and Primary analyses described in Substudy 2 Protocol Amendment 4 Section 10.5 will not be conducted, only the Final Analysis will be undertaken. 3) No subgroup analyses will be undertaken as a result of recruiting fewer participants than the planned target sample size.

# 1.1. Objectives, Estimands, and Endpoints

The full list of objectives and endpoints below is the list given in the Substudy 2 Protocol Amendment 4.

As of Substudy 2 SAP Amendment 1: Due to early termination of this substudy, only a subset of the exploratory endpoints will be analysed.

# 1.1.1. Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| To assess the safety, tolerability and determine recommended phase 2 dose (RP2D) of GSK3845097 in HLA-A*02:01, HLA-A*02:05 | Frequency of dose-limiting toxicities (DLTs) |
| and/or HLA-A*02:06 positive participants with NY-ESO-1 and/or LAGE-1a positive, previously treated, advanced (metastatic or unresectable) | <ul> <li>Frequency and severity of adverse<br/>events (AEs), serious adverse events<br/>(SAEs) and AEs of special interest</li> </ul> |
| SS and MRCLS | (AESI; as defined in the core protocol) |
| Secondary – Efficacy | |
| To investigate the anti-tumor activity of GSK3845097 in HLA-A*02:01, HLA-A*02:05 and/or HLA-A*02:06 positive participants with | Overall Response Rate (ORR) (investigator assessed according to RECIST v1.1) |
| NY-ESO-1 and/or LAGE-1a positive, previously treated, advanced (metastatic or unresectable) SS and MRCLS | Duration of Response (DoR) |
| Secondary – Pharmacokinetics (PK) | |
| To characterize in vivo cellular PK profile (levels, | Maximum transgene expansion (Cmax) |
| expansion, persistence) of GSK3845097 over time | Time to Cmax (Tmax) |

| Objectives | Endpoints |
|---|---|
| | Area under the time curve from zero to<br>time t AUC(0-t), as data permit |
| Exploratory | |
| CCI | |
| _ | |
| - | |
| - | |



# 1.2. Study Design



EOT = end of treatment (i.e., interventional) portion of the trial; HLA = human leukocyte antigen; ICF = informed consent form; LTFU = long-term follow-up; MRCLS = myxoid/round cell liposarcoma; SS = synovial sarcoma.

- 1. Screening, including HLA typing and antigen testing, may be done in this study or as part of a separate Pre-screening protocol.
- 2. Sponsor will inform Investigators of the participant assignments between substudies and indicate if the participant is a sentinel participant and the number of remaining slots.
- 3. The first participant to be dosed will receive the total dose in 2 separate infusions as aliquots of ~30% and ~70% of the total manufactured dose, administered 7 days apart. The second infusion will only be administered if no acute toxicities preventing full dosing are observed. If no DLTs are reported for the participants receiving split doses, then all subsequent participants administered the particular product will receive the full dose as a single i.e., one-time, infusion.
- 4. See Section 5.3.1 of this substudy Protocol for definition of the end of interventional phase for a participant.
- 5. The LTFU assessments and procedures may be done in this study or under a separate LTFU protocol.

#### **Dose Confirmation Phase LTFU** Dose Expansion Phase @ RP2D Dose Confirmation Phase in SS/MRCLS Progressive disease after SOC treatment No brain metastasis allowed Dose Expansion Phase @RP2D in SS/MRCLS Disease confirmed by translocation Measurable disease N=10 total evaluable participants @ RP2D LTFU for total Supportive chemotherapy permitted Followed until PD or the end of interventional phase, whichever of 15 years between screening and lymphodepletion is sooner Split dose for sentinel participant 2-week staggering for first 3 participants Potential Dose de-escalation Safety review after each 3 dosed

LTFU = long-term follow-up; MRCLS = myxoid/round cell liposarcoma; PD = progressive disease; RP2D = recommended phase 2 dose; SS = synovial sarcoma.

# Design Features

- This is a first time in human (FTIH) non-randomized, open-label substudy to investigate GSK3845097 in previously treated participants with advanced (metastatic or unresectable) synovial sarcoma (SS) and myxoid/round cell liposarcoma (MRCLS). This substudy will consist of two phases: Dose Confirmation Phase and Dose Expansion Phase.
- Dose Confirmation Phase (n=6-15)

### **Overview of Study Design and Key Features**

- The primary objective of the dose confirmation phase is to identify the RP2D of GSK3845097. RP2D will be determined as the maximum tolerated dose (MTD) or lower that provides adequate biologic activity with superior tolerability. The MTD is defined as the dose that maximizes the probability of target toxicity of 30% while controlling the probability of excessive or unacceptable toxicity
- To find the RP2D, modified toxicity probability interval 2 (mTPI-2) design will be implemented. Participants will be recruited and treated in blocks of three. The design aims to identify a dose with a true underlying toxicity rate of 30, with a range of 25% to 35%.
- The dose will be re-escalated/de-escalated based on all available data. The DLT information on all participants enrolled in the trial is used to update the estimated dose toxicity relationship and provide supportive information in addition to the mTPI-2 design in the next re-escalation/de-escalation decision.
- Dose Selection Committee (DSC) will meet after the DLT period in every 3 participants to enable dose decision until the final dose selection is achieved (6 to 15 participants).
- The final determination of RP2D will be based on the mTPI-2 recommended dose, as defined as ≥6 participants treated at this dose and an observed toxicity rate closest to the targeted toxicity rate at 30% after isotonic regression, in addition to considering the clinical response rate and available PK and PD data generated from all participants.

### • Dose Expansion Phase (n = 10)

- After RP2D has been determined, the cohort will enroll additional participants to ensure n=10 participants have become evaluable at the RP2D.
- Evaluable participants are those who have received T-cell infusion and have completed at least 2 post-baseline disease assessments since infusion or have progressed or died or were withdrawn from the substudy.
- For each individual participant, the study will consist of the following: 1) Screening, 2) Leukapheresis and manufacture, 3) Interventional Phase (Lymphodepletion, Treatment and Follow-up), 4) Long-term follow-up (LTFU). Part 1: Screening Target expression screening for the presence of HLA- A\*02:01, HLA-A\*02:05 and/or HLA-A\*02:06 positivity and tumour expression of NY-ESO-1 and/or LAGE-1a, leukapheresis eligibility screening within 28 days prior to the day of the scheduled leukapheresis procedure. Part 2: Leukapheresis and Manufacture Eligible participants, upon study enrollment, will undergo leukapheresis. The initiation of leukapheresis procedure constitutes enrollment in the study. The collected T cells will be sent for manufacturing. Part 3: Interventional Phase (Lymphodepletion, Treatment and Follow-up) Treatment fitness assessment and eligibility confirmation, Lymphodepletion from Days -7 to -4, GSK3845097 intravenous (IV) infusion on Day 1 and follow-up until the end of study (as defined in Protocol Section 5.3 of this Substudy). Part 4: Long-Term Follow-Up (LTFU) Long-term follow-up phase for up to 15 years from the date of GSK3845097 infusion.

# Study intervention

### Leukapheresis

 Participants will undergo leukapheresis to obtain starting material for the manufacture of GSK3845097.

#### Bridging therapy and/or standard of care intermediate anti-cancer therapy

 Bridging or standard of care systemic chemotherapy, experimental therapy and/or local therapy (e.g., radiotherapy, cryoablation, surgical resection) may be administered between Target Expression Screening and Leukapheresis.



| Overview of Study Design and Key Features | |
|---|---|
| | An interim analysis will be performed for each cohort after 10 participants in the cohort<br>are evaluable at the RP2D. These analyses may be performed earlier with fewer than 10<br>evaluable participants at the RP2D if it is clear from the accumulated data what the<br>decision at 10 evaluable participants treated at RP2D would be. In the event that an<br>early futility decision is made for ORR then enrollment to the cohort will be closed. |
| | Primary Analysis The primary analysis for each cohort will be performed after enrollment to the cohort is complete and all the enrolled participants in the cohort that will receive T-cell infusion |
| | have done so and of those: at least 80% have confirmed disease progression or died, or were withdrawn or lost to follow-up from the substudy; and all the remaining infused participants have completed at least 2 post baseline disease assessments since infusion. |
| | <ul> <li>If the primary analysis for a cohort is expected to occur within 9 months of the final<br/>analyses for the cohort, then the primary analysis may be omitted and only the final<br/>analyses carried out.</li> </ul> |
| Time & Events | For the schedule of activities refer to Section 2 of the substudy Protocol. |

# 2. STATISTICAL HYPOTHESES

The primary aim is to determine the recommended phase 2 dose, safety profiles and pharmacology of GSK3845097. Descriptive methods will be used in analyses of the data from this substudy. No inferential statistical hypothesis testing will be conducted.

The null hypothesis for the secondary endpoint ORR is: p=40%

The alternative hypothesis is: p=60%

The assumptions for the secondary endpoint of ORR, as defined in the core SAP Section 4.3.1.1.1, underlying the design are detailed below:

The null hypothesis for the secondary endpoint ORR is: p=40%

The alternative hypothesis is: p=60%

# 2.1. Multiplicity Adjustment

No formal statistical hypothesis testing will be performed and therefore no multiplicity adjustment is required.

# 3. ANALYSIS SETS

Refer to Section 3 of the core SAP.

### 4. STATISTICAL ANALYSES

### 4.1. General Considerations

# 4.1.1. General Methodology

No inferential statistical hypothesis testing will be conducted, i.e., no p-values will be calculated. Unless otherwise specified, continuous data will be summarized using descriptive statistics: number of subjects (n), mean, standard deviation, median, minimum, and maximum. Categorical data will be summarized as the number and percentage of participants in each category.

Confidence intervals will use 95% confidence levels unless otherwise specified.

For safety, data will be summarised by phase. In general, safety data will be displayed by actual dose received (total number of transduced T-cells) using the following columns: 0.1-0.8 x 10^9 vs. 1-8 x 10^9 (mITT population tables). Please refer to Table 1 in the core SAP for the applicable tables that are to be displayed by the planned dose. The planned dose tables will use the following columns: DL-1 (for 0.1-0.8 x 10^9) and DL1 (for 1-8 x 10^9). For tables on the ITT population, an additional column of "No treatment" will be included consisting of those who did not receive lymphodepletion chemotherapy and T-cell infusion.

For efficacy, data will be summarised by phase. The planned analyses will only include the efficacy data from the cohort of interest for the analyses. Data will be displayed by actual dose received (total number of transduced T-cells) using the following columns: 0.1-0.8 x 10<sup>9</sup> vs. 1-8 x 10<sup>9</sup> (mITT population tables only)

Details of the planned displays are provided in the core and Substudy 2 Output and Programming Specification (OPS) and are based on GSK data standards and statistical principles.

#### 4.1.2. Baseline Definition

Refer to Section 4.1.2. of the core SAP.

# 4.2. Primary Endpoint(s) Analyses

Refer to Section 4.2. of the core SAP.

# 4.3. Secondary Endpoint(s) Analyses

Refer to Section 4.3. of the core SAP.

# 4.4. Exploratory Endpoint(s) Analyses

Refer to Section 4.4. of the core SAP.

# 4.5. Safety Analyses

Refer to Section 4.5. of the core SAP.

# 4.6. Other Analyses

## 4.6.1. Subgroup analyses

Due to early termination of this substudy, subgroup analyses will not be conducted.

# 4.7. Interim Analyses

Protocol-planned analyses include an Interim, Primary and Final analysis. However, due to the early termination of all substudies, only a final analysis will be conducted.

#### 4.7.1. Dose Confirmation Phase

As of Substudy 2 SAP Amendment 1: Note that this substudy was terminated prior to the determination of RP2D, and so there will be no RP2D recommended based on the mTPI-2.

For the dose confirmation phase there are no formal interim analyses planned.

All available safety and tolerability data including safety laboratory data, end and PK data (if applicable) and the safety profile observed will be reviewed during the DSC meetings to inform dose escalation decisions and support the RP2D decision. The DSC meetings will occur after the DLT period (28 days after last IP dose) in every 3 participants to enable dose decision until the final dose selection is achieved.

The DLT information on all participants enrolled in the trial is used to update the estimated dose toxicity relationship and provide supportive information in addition to the mTPI-2 (Section 4.7.1.1) in the next re-escalation/de-escalation decision; the mTPI-2 approach is expected to be used as the primary criteria for dose escalation.

The final determination of RP2D will be based on the mTPI-2 (Section 4.7.1.1) recommended dose, as defined as ≥6 participants treated at this dose and an observed toxicity rate closest to the targeted toxicity rate at 30% after isotonic regression, in addition to considering the clinical response rate and available PK and Pharmacodynamics data generated from all participants.

### 4.7.1.1. Modified Toxicity Probability Interval 2 (mTPI-2) Design

As of Substudy 2 SAP Amendment 1: Note that this substudy was terminated prior to the determination of RP2D, and so there will be no RP2D recommended based on the mTPI-2.

The dose confirmation phase of this study is based on mTPI-2 [Guo, 2017] design. mTPI-2 is implemented within a formal Bayesian decision framework. The mTPI-2 design for this study assumes the underlying toxicity rate for maximum tolerated dose of

GSK3845097 falls within the range from 25% to 35% and is centred at 30%. The stopping rule threshold for excessive toxicity is 0.95 and the prior probability of toxicity at each dose is distributed as Beta(1,1).

The monitoring rules guiding dose escalation are provided in Table 1. Columns provide the numbers of participants treated at the current dose level, and rows provide the corresponding numbers of participants experiencing DLTs. The entries of the table are dose-finding decisions (i.e., R, S, and D) representing re-escalating the dose, staying at the same dose, and de-escalating the dose. In addition, decision U means that the current dose level is unacceptable because of high toxicity and should be excluded from the trial. For example, when one of three participants experiences toxicity, the decision can be located at row 1 and column 3, which is S—to stay at the current dose level. Consequently, the next block of participants will be treated at the same dose level currently being used. If zero of three participants experience toxicity, the decision is at row 0 and column 3, which is R—to re-escalate. Thus, the next block of participants will be treated at the higher dose level, if available. If three of three participants experience toxicity, the decision is to de-escalate to the lower dose level and exclude the current dose from the trial, because the toxicity level is unacceptable.

The final determination of RP2D will be based on the mTPI-2 recommended dose, as defined as ≥6 participants treated at this dose and an observed toxicity rate closest to the targeted toxicity rate at 30% after isotonic regression, in addition to considering the clinical response rate and available PK and PD data generated from all participants.

Table 1 DLT De-escalation/Re-Escalation Rules

| 50 | | 3 | 6 | 9 | 12 | 15 |
|---|---|---|---|---|---|---|
| ling. | 0 | R | R | R | R | R |
| mit | 1 | S | R | R | R | R |
| [r] | 2 | D | S | R | R | R |
| se | 3 | U | D | S | S | R |
| DC<br>S) | 4 | | U | D | S | S |
| narticipants with Do<br>Toxicities (DLTs)<br>at the current dose | 5 | | U | U | D | S |
| (D) ent | 6 | | U | U | D | D |
| ies<br>ies | 7 | | | U | U | D |
| ipa<br>citi | 8 | | | U | U | U |
| tic<br>oxi<br>the | 9 | | | U | U | U |
| Dar<br>T | 10 | | | | U | U |
| | 11 | | | | U | U |
| Number of participants with Dose Limiting<br>Toxicities (DLTs)<br>at the current dose | 12 | | | | U | U |
| l qu | 13 | | | | | U |
| E | 14 | | | | | U |
| | 15 | | | | | U |

R=Re-escalate to the higher dose if applicable OR Stay at the current dose otherwise

D=De-escalate to the lower dose if applicable OR Stay at the current dose otherwise

Target toxicity level=30%

e1=e2=0.05

S=Stay at the current dose

U=The current dose is unacceptably toxic

### 4.7.2. Dose Expansion Phase

As of Substudy 2 SAP Amendment 1: Note that this substudy was terminated prior to the determination of RP2D. Hence this section of text is no longer applicable.

An interim analysis for futility will be performed for each cohort after 10 participants in the cohort are evaluable at the RP2D. Evaluable subjects who received RP2D in the dose confirmation phase will be included in the 10 participants. The endpoint assessed for futility is the Overall Response Rate (ORR), defined as the proportion of participants with an investigator-assessed confirmed complete response (CR) or confirmed partial response (PR) per RECIST v1.1. The endpoint assessed for futility is the Overall Response Rate (ORR), defined as the proportion of participants with an investigator-assessed confirmed complete response (CR) or confirmed partial response (PR) per RECIST v1.1.

The interim analysis may be performed earlier with fewer than 10 evaluable participants at the RP2D if it is clear from the accumulated data what the decision at 10 evaluable participants treated at RP2D would be.

Futility rules are provided in Table 2 and justification for these rules is provided in Section 5. Note that these rules are for guidance only and futility decisions will be made based on the totality of the data. In the event that an early futility decision is made then enrollment to the cohort will be closed.

If there are 4 or fewer responders out of 10 evaluable participants, then the substudy may stop for futility (see Section 5 for justification). This interim analysis may be performed earlier with less than 10 evaluable participants at the RP2D if it is clear from the accumulated data what the decision at 10 evaluable participants treated at RP2D would be (Table 2). For example, if no responders are observed in the first 6 evaluable participants at the RP2D then an early interim analysis may be conducted.

Table 2 Interim Analysis Futility Rules

| Interim A | Analysis | Early Interim Analysis | |
|---|---|---|---|
| Number of participants | Stop for futility if no. of | Number of participants | Stop for futility if no. of |
| evaluable at RP2D | responders is | evaluable at RP2D | responders is |
| 10 | ≤4 | 6 | 0 |

Abbreviations: RP2D = Recommended Phase 2 Dose.

Criteria are for guidance only. Final decisions will be based on a review of the totality of the data.

# 4.7.3. Primary Analysis

As of Substudy 2 SAP Amendment 1: Protocol-planned analyses include an Interim, Primary and Final analysis. However, due to the early termination of all substudies, only a final analysis will be conducted.

Refer to Section 4.7.2 in the core SAP and Section 10.5.1.1 in the Substudy 2 Protocol.

# 4.7.4. Final Analysis

Refer to Section 4.7.3 in the core SAP.

# 4.8. Changes to Protocol Defined Analyses

Any changes from the originally planned statistical analysis specified in the protocol amendment 4 (Dated: 27-May-2022) are described in the Core SAP Section 4.8.

# 5. SAMPLE SIZE DETERMINATION

The Dose Confirmation phase would need 6-15 participants to establish RP2D (see mTPI-2 simulation results in core SAP Section 6.4.1). Thus, the total expected maximal number of participants in the Dose Confirmation phase is 15.

Once the RP2D has been established, the substudy will expand to up to n=10 evaluable participants treated at that dose. The null hypothesis is that the true ORR is 40% and the alternative hypothesis is that the true ORR is 60%. This substudy size was chosen to allow for early stopping of further development due to futility if the posterior probability that the ORR is less than 60% is >90%. This is equivalent to observing 4 or fewer responders out of 10 treated participants. It was assumed that the prior distribution for the response rate follows an uninformative Beta(a=0.02, b=0.08) distribution. Additionally, if the true ORR is 40%, the probability of observing 4 or fewer responders out of 10 treated participants is 63% and if the true ORR is 60% the probability of observing 4 or fewer responders out of 10 treated participants is 17%. These decision rules are for guidance only and the final decision for stop for futility will be determined based on the totality of the data.

If supported by safety and efficacy results, additional participants may be enrolled to confirm the safety and efficacy via a protocol amendment or as part of a separate protocol.

• For this substudy, five or more confirmed responses (CR or PR) out of 10 evaluable participants treated at RP2D may provide sufficient efficacy evidence to expand and enroll additional participants.

This will serve as guidance for final decisions regarding enrollment of additional participants, which will be based on a review of the totality of the data.

# 6. SUPPORTING DOCUMENTATION

Refer to Section 6 of the core SAP. Any differences or additional analyses are specified below.

# 6.1. Appendix 1 Study Population Analyses

# 6.1.1. Demographic and Baseline Characteristics

Disease characteristics at initial diagnosis and screening will be analysed as per Section 6.1.2 in the core SAP. Presentations will also include the specific disease characteristics related to SS and MRCLS that are entered on separate corresponding eCRF pages. For SS this will include the extent of the disease at screening (local unresectable or metastatic), SYT-SSX translocation (SYT-SSX1, SYT-SSX2, SYT-SSX4 or not applicable or other) and histology type (monophasic, biphasic, not available, or other). For MRCLS this will include the extent of disease at screening (local unresectable or metastatic), specific translocation (FUS-DDIT3, EWSR1-DDIT3, not applicable or other) and percent round cell.

# 7. REFERENCES

Guo Wang SJ, Yang S, Lynn H, Ji Y. A Bayesian interval dose-finding design addressing Ockham's razor: mTPI-2. Contemp Clin Trials. 2017; 58:23-33.